CLINICAL TRIAL: NCT06615258
Title: Investigation of the Effect of Breathing-based Pelvic Floor Muscle Training on Menstrual Symptoms, Pain and Quality of Life in Women With Primary Dysmenorrhea: A Randomized-Controlled Trial
Brief Title: The Effect of Breathing-based Pelvic Floor Muscle Training on Menstrual Symptoms, Pain and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Assistant Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYY_3
Record Dates: First submitted 2024-09-12; First posted 2024-09-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Dysmenorrhea Primary; Pain Management; Diaphragmatic Breathing; Pelvic Floor Muscle Exercise
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DNS Based breathing exercises+PFMT (Experimental): Dynamic Neuromuscular Stabilization (DNS)-based respiratory training and pelvic floor muscle training (PFMT) will be applied.
  Interventions: Behavioral: Dynamic Neuromuscular Stabilization based breathing training and pelvic floor muscle training
- PFMT (Active Comparator): Pelvic floor muscle training (PFMT) will be applied.
  Interventions: Behavioral: Pelvic floor muscle training
- Control Group (No Intervention): No intervention will be made to the participants in this group.

INTERVENTIONS:
Behavioral: Dynamic Neuromuscular Stabilization based breathing training and pelvic floor muscle training — DNS-based breathing exercises will be taught to the women in this group using tactile biofeedback. To create tactile stimulation, one of the hard sponges placed within a belt will be positioned anteriorly in the inguinal region, and the other posteriorly in the Grynfeltt-Lesshaft triangle region. Breathing training will be provided in 3 different positions: sitting, crawling, and happy baby pose.
  Pelvic floor muscle training: PFME will consist of 2 parts: relaxation training for pelvic floor muscles and pelvic floor muscle exercises.
  Pelvic floor muscles will be given relaxation training in 3 different relaxation positions (modified butterfly pose, child pose and deep squatting position) suggested by Çeliker Tosun et al. PFME will be taught by the physiotherapist in the side-lying with external coccyx palpation. PFME will be applied in the hook-lying position, sitting position and standing position.
  Arms: DNS Based breathing exercises+PFMT
Behavioral: Pelvic floor muscle training — Pelvic floor muscle training: PFME will consist of 2 parts: relaxation training for pelvic floor muscles and pelvic floor muscle exercises. Pelvic floor muscles will be given relaxation training in 3 different relaxation positions (modified butterfly pose, child pose and deep squatting position) suggested by Çeliker Tosun et al. PFME will be taught by the physiotherapist in the side-lying with external coccyx palpation. PFME will be applied in the hook-lying position, sitting position and standing position.
  Arms: PFMT

SUMMARY:
Primary dysmenorrheic (PD) pain usually begins during adolescence, at menarche or shortly after (6-24 months), and has a clear and predictable temporal pattern. The pain typically radiates to the back and thighs and lasts for 8-72 hours. The pain is most severe on the first and/or second day of menstrual bleeding. Additionally, systemic symptoms such as nausea, vomiting, diarrhea, fatigue, and insomnia often accompany the pain. In secondary dysmenorrhea, it can result from a range of identifiable pathological conditions, including endometriosis, adenomyosis, fibroids, and pelvic inflammatory disease. Other gynecological symptoms such as intermenstrual bleeding and menorrhagia may also accompany it, depending on the underlying condition. Empirical treatment approaches have been reported as appropriate for patients with primary dysmenorrhea based on symptoms and physical examination results. Recent studies have indicated that during diaphragmatic breathing, all the muscles that make up the thoracic and abdominal walls should expand in a cylindrical manner in all directions through synchronized eccentric activity. Thus, a more effective result will occur with the concentric contraction and 360-degree expansion of the diaphragm during inspiration, which raises intra-abdominal pressure .

Within the framework of this information, the aim of this study is to examine the effects of respiration-based physiotherapy approaches on menstrual symptoms, pain, and quality of life in women with PD.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35,
* Voluntary participation,
* Having a regular menstrual cycle (every 24-35 days) ,
* Menstrual pain intensity of 3/10 or higher on the Visual Analog Scale during the initial assessment,
* Pain radiating to the back, legs, lower abdominal, or suprapubic region during menstruation,
* Restriction of daily living activities due to pain,
* Requirement for medical intervention or self-medication to control the pain.

Exclusion Criteria:

* History of pelvic pathology and/or surgery that could cause pain,
* Neurological or psychological disorders,
* Anovulation,
* Other diseases that could affect chest expansion or the respiratory system (COPD, asthma, pneumonia, bronchiectasis, etc.),
* Being pregnant, having a positive birth control status, or being less than 6 months postpartum,
* Use of an intrauterine device,
* History of childbirth or miscarriage. Individuals who miss two consecutive exercise sessions will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change of Menstruation Symptom Scale score | 4 weeks after the intervention
  Individuals menstrual pain and symptoms will be assessed with the Menstruation Symptom Scale. The Turkish validity and reliability of this scale was conducted by Güvenç et al. in 2014. The MSS is a five-point Likert-type scale consisting of twenty-two items. Participants are asked to give a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. The scale has three sub-dimensions: 'Negative Effects/Somatic Complaints' (Items 1-13), 'Menstrual Pain Symptoms' (Items 14-19) and 'Coping Methods' (Items 20-22). The highest score that can be obtained from the scale is 110, the lowest score is 22.
Change in the McGill pain questionnaire score | 4 weeks after the intervention
  The McGill pain questionnaire will be used to assess the severity and quality of menstrual pain in individuals. This questionnaire consists of 11 words to determine the sensory aspect of pain and 4 words to determine the affective aspect, totaling 15 different words related to the quality of pain. In addition, the pain intensity felt at the time of measurement is measured with VAS, and the total pain intensity evaluated is measured with a 6-point Likert-type scale.

SECONDARY OUTCOMES:
Change of Menstruation Symptom Scale score | 3 months after the intervention
  Individuals menstrual pain and symptoms will be assessed with the Menstruation Symptom Scale. The Turkish validity and reliability of this scale was conducted by Güvenç et al. in 2014. The MSS is a five-point Likert-type scale consisting of twenty-two items. Participants are asked to give a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. The scale has three sub-dimensions: 'Negative Effects/Somatic Complaints' (Items 1-13), 'Menstrual Pain Symptoms' (Items 14-19) and 'Coping Methods' (Items 20-22). The highest score that can be obtained from the scale is 110, the lowest score is 22.
Change of Quality of Life score | 4 weeks after the intervention
  Short Form-36 is a 36-question self-assessment scale consisting of eight subscales. This scale consists of physical function (10 items), role limitations (physical (4 items) and emotional problems (3 items), pain (2 items), vitality (4 items), social function (2 items), mental health (5 items) and general health (5 items) subscales. Each subscale is scored between 0-100, with "0" indicating the lowest and "100" indicating the best quality of life level.
Change in the McGill pain questionnaire score | 3 months after the intervention
  The McGill pain questionnaire will be used to assess the severity and quality of menstrual pain in individuals. This questionnaire consists of 11 words to determine the sensory aspect of pain and 4 words to determine the affective aspect, totaling 15 different words related to the quality of pain. In addition, the pain intensity felt at the time of measurement is measured with VAS, and the total pain intensity evaluated is measured with a 6-point Likert-type scale.
Change of Quality of Life score | 3 months after the intervention
  Short Form-36 is a 36-question self-assessment scale consisting of eight subscales. This scale consists of physical function (10 items), role limitations (physical (4 items) and emotional problems (3 items), pain (2 items), vitality (4 items), social function (2 items), mental health (5 items) and general health (5 items) subscales. Each subscale is scored between 0-100, with "0" indicating the lowest and "100" indicating the best quality of life level.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir University of Economics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No